CLINICAL TRIAL: NCT01627249
Title: A Comparative Effectiveness Study of Intravitreal Aflibercept, Bevacizumab and Ranibizumab for Diabetic Macular Edema
Brief Title: Comparative Effectiveness Study of Intravitreal Aflibercept, Bevacizumab, and Ranibizumab for Diabetic Macular Edema
Acronym: Protocol T
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Eye Institute (NEI) (NIH); Genentech, Inc. (Industry); Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DRCR.net Protocol T; EY14231 (Other Grant/Funding Number: National Eye Institute); EY23207 (Other Grant/Funding Number: National Eye Institute); EY18817 (Other Grant/Funding Number: National Eye Institute)
Record Dates: First submitted 2012-06-21; First posted 2012-06-25 (Estimated); Results first posted 2015-12-16 (Estimated); Last update posted 2020-08-10 (Actual); Status verified 2020-07

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic Macular Edema; anti-vascular endothelial growth factor

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ranibizumab (Active Comparator)
  Interventions: Drug: 0.3 mg intravitreal ranibizumab
- Aflibercept (Experimental)
  Interventions: Drug: 2.0 mg intravitreal aflibercept
- Bevacizumab (Experimental)
  Interventions: Drug: 1.25 mg intravitreal bevacizumab

INTERVENTIONS:
Drug: 2.0 mg intravitreal aflibercept — Intravitreal injection of 2.0 mg aflibercept at baseline and up to every 4 weeks using defined retreatment criteria.
  Arms: Aflibercept
Drug: 1.25 mg intravitreal bevacizumab — Intravitreal injection of 1.25 mg bevacizumab at baseline and up to every 4 weeks using defined retreatment criteria.
  Arms: Bevacizumab
Drug: 0.3 mg intravitreal ranibizumab — Intravitreal injection of 0.3 mg ranibizumab (Lucentis™) at baseline and up to every 4 weeks using defined retreatment criteria.
  Arms: Ranibizumab

SUMMARY:
Although multiple studies have suggested that treatment with ranibizumab is safe and efficacious and superior to focal/grid laser alone for patients with center-involved diabetic macular edema (DME), there may be barriers in place to widespread adoption of ranibizumab use given its high cost per dose and the need for multiple treatments over time. Prioritizing resources from a public health policy perspective could be easier if more precise estimates regarding the risks and benefits of other anti-vascular endothelial growth factor (anti-VEGF) therapies were available, especially when the difference in costs could be billions of dollars over just a few years. Thus, there is a clear rationale at this time to explore potential anti-VEGF alternatives to ranibizumab that might prove to be as or more efficacious, might deliver equally lasting or longer-lasting treatment effects, and cost substantially less. Of the potentially available alternative anti-VEGF agents for this trial, bevacizumab and aflibercept are the best candidates for a direct comparison study. Bevacizumab shares the most similar molecular structure, costs far less, and is widely available. Furthermore, there is already preliminary evidence to suggest that it may be efficacious in the treatment of DME and it is already being widely used for this indication. Although aflibercept has a similar cost per unit dose to ranibizumab, it has the potential to decrease treatment burden and associated cost. If results from a comparative trial demonstrate improved efficacy or suggest similar efficacy of bevacizumab or aflibercept over ranibizumab, this information might give clinicians scientific rationale to substitute either one of these drugs for ranibizumab in the treatment of DME, and might thereby have substantial implications for public policy in terms of future estimates of health care dollars and possibly number of treatments necessary for anti-VEGF treatment of diabetic macular disease.

Because of its availability and lower cost, bevacizumab is already currently in widespread clinical use for treatment of DME despite the lack of FDA approval for this indication. Thus, a clinical trial that suggested whether bevacizumab could be used as a safe and efficacious alternative to ranibizumab could substantially impact nationwide practice patterns for treatment of DME by either validating the current use of bevacizumab or by demonstrating improved outcomes with ranibizumab or aflibercept treatment for DME.

Study Objective The primary objective of the proposed research is to compare the efficacy and safety of (1) intravitreal aflibercept, (2) intravitreal bevacizumab, and (3) intravitreal ranibizumab when given to treat central-involved DME in eyes with visual acuity of 20/32 to 20/320.

DETAILED DESCRIPTION:
A five year follow-up visit is being conducted to gather information on long term outcomes

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Individuals <18 years old are not being included because DME is so rare in this age group that the diagnosis of DME may be questionable.
* Diagnosis of diabetes mellitus (type 1 or type 2)
* Any one of the following will be considered to be sufficient evidence that diabetes is present:
* Current regular use of insulin for the treatment of diabetes
* Current regular use of oral anti-hyperglycemia agents for the treatment of diabetes
* Documented diabetes by American Diabetes Association and/or World Health Organization criteria (see Procedures Manual for definitions)
* At least one eye meets the following study eye criteria:

  * Best corrected Electronic-Early Treatment Diabetic Retinopathy Study visual acuity letter score ≤ 78 (i.e., 20/32 or worse) and ≥ 24 (i.e., 20/320 or better) within eight days of randomization.
  * On clinical exam, definite retinal thickening due to diabetic macular edema involving the center of the macula.
  * Diabetic macular edema present on optical coherence tomography (OCT) (central subfield thickness on OCT >250 µm on Zeiss Stratus or the equivalent on spectral domain OCTs based on gender specific cutoffs), within eight days of randomization.
  * Investigator must verify accuracy of OCT scan by ensuring it is centered and of adequate quality (for Zeiss Stratus, standard deviation of center point thickness should be ≤ 10% of the center point thickness and signal strength should be ≥ 6)
  * Media clarity, pupillary dilation, and individual cooperation sufficient for adequate fundus photographs
* Able and willing to provide informed consent.

Exclusion Criteria:

* Significant renal disease, defined as a history of chronic renal failure requiring dialysis or kidney transplant.
* A condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure, cardiovascular disease, and glycemic control).

  •Individuals in poor glycemic control who, within the last four months, initiated intensive insulin treatment (a pump or multiple daily injections) or plan to do so in the next four months should not be enrolled.
* Participation in an investigational trial within 30 days of randomization that involved treatment with any drug that has not received regulatory approval for the indication being studied at the time of study entry.

  • Note: study participants cannot receive another investigational drug while participating in the study.
* Known allergy to any component of the study drug.
* Blood pressure > 180/110 (systolic above 180 OR diastolic above 110).

  • If blood pressure is brought below 180/110 by anti-hypertensive treatment, individual can become eligible.
* Myocardial infarction, other acute cardiac event requiring hospitalization, stroke, transient ischemic attack, or treatment for acute congestive heart failure within 4 months prior to randomization.
* Systemic anti-VEGF or pro-VEGF treatment within four months prior to randomization or anticipated use during the study.

  • These drugs cannot be used during the study.
* For women of child-bearing potential: pregnant or lactating or intending to become pregnant within the next 24 months.
* Women who are potential study participants should be questioned about the potential for pregnancy. Investigator judgment is used to determine when a pregnancy test is needed.
* Individual is expecting to move out of the area of the clinical center to an area not covered by another clinical center during the first 12 months of the study.

The following exclusions apply to the study eye only (i.e., they may be present for the nonstudy eye):

* Macular edema is considered to be due to a cause other than diabetic macular edema.
* An eye should not be considered eligible if: (1) the macular edema is considered to be related to ocular surgery such as cataract extraction or (2) clinical exam and/or OCT suggest that vitreoretinal interface abnormalities (e.g., a taut posterior hyaloid or epiretinal membrane) are the primary cause of the macular edema.
* An ocular condition is present such that, in the opinion of the investigator, visual acuity loss would not improve from resolution of macular edema (e.g., foveal atrophy, pigment abnormalities, dense subfoveal hard exudates, nonretinal condition).
* An ocular condition is present (other than diabetes) that, in the opinion of the investigator, might affect macular edema or alter visual acuity during the course of the study (e.g., vein occlusion, uveitis or other ocular inflammatory disease, neovascular glaucoma, etc.).
* Substantial cataract that, in the opinion of the investigator, is likely to be decreasing visual acuity by three lines or more (i.e., cataract would be reducing acuity to 20/40 or worse if eye was otherwise normal).
* History of an anti-VEGF treatment for DME in the past 12 months or history of any other treatment for DME at any time in the past four months (such as focal/grid macular photocoagulation, intravitreal or peribulbar corticosteroids).
* Enrollment will be limited to a maximum of 25% of the planned sample size with any history of anti-VEGF treatment for DME. Once this number of eyes has been enrolled, any history of anti-VEGF treatment for DME will be an exclusion criterion.
* History of pan-retinal photocoagulation within four months prior to randomization or anticipated need for pan-retinal photocoagulation in the six months following randomization.
* History of anti-VEGF treatment for a disease other than DME in the past 12 months.
* History of major ocular surgery (including vitrectomy, cataract extraction, scleral buckle, any intraocular surgery, etc.) within prior four months or anticipated within the next six months following randomization.
* History of YAG capsulotomy performed within two months prior to randomization.
* Aphakia.
* Exam evidence of external ocular infection, including conjunctivitis, chalazion, or significant blepharitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Actual)
Dates: Start 2012-08; Primary Completion 2014-10 (Actual); Study Completion 2019-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John A Wells, MD, Study Chair — Palmetto Retina Center
Locations (90):
- United States (90):
  - Retina Associates, Tucson, Arizona
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Loma Linda University Health Care, Dept. of Ophthalmology, Loma Linda, California
  - Southern California Desert Retina Consultants, MC, Palm Desert, California
  - California Retina Consultants, Santa Barbara, California
  - Bay Area Retina Associates, Walnut Creek, California
  - Retinal Consultants of Southern California Medical Group, Inc., Westlake Village, California
  - New England Retina Associates, Norwich, Connecticut
  - Gulf Coast Retina Center, Clearwater, Florida
  - Retina Group of Florida, Fort Lauderdale, Florida
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - Central Florida Retina Institute, Lakeland, Florida
  - Ocala Eye Retina Consultants, Ocala, Florida
  - Magruder Eye Institute, Orlando, Florida
  - Fort Lauderdale Eye Institute, Plantation, Florida
  - Sarasota Retina Institute, Sarasota, Florida
  - Retina Associates of Florida, P.A., Tampa, Florida
  - Emory Eye Center, Atlanta, Georgia
  - Georgia Retina, P.C., Atlanta, Georgia
  - Thomas Eye Group, Atlanta, Georgia
  - Southeast Retina Center, P.C., Augusta, Georgia
  - Retina Consultants of Hawaii, Inc., Honolulu, Hawaii
  - Northwestern Medical Faculty Foundation, Chicago, Illinois
  - University of Illinois at Chicago Medical Center, Chicago, Illinois
  - NorthShore University HealthSystem, Glenview, Illinois
  - Raj K. Maturi, M.D., P.C., Indianapolis, Indiana
  - John-Kenyon American Eye Institute, New Albany, Indiana
  - Medical Associates Clinic, P.C., Dubuque, Iowa
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - Retina Associates, P.A., Shawnee Mission, Kansas
  - Retina and Vitreous Associates of Kentucky, Lexington, Kentucky
  - Paducah Retinal Center, Paducah, Kentucky
  - Elman Retina Group, P.A., Baltimore, Maryland
  - Wilmer Eye Institute at Johns Hopkins, Baltimore, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Joslin Diabetes Center, Boston, Massachusetts
  - Vitreo-Retinal Associates, PC, Worcester, Massachusetts
  - Henry Ford Health System, Dept of Ophthalmology and Eye Care Services, Detroit, Michigan
  - Retina Vitrous Center, Grand Blanc, Michigan
  - Retina Specialists of Michigan, Grand Rapids, Michigan
  - Vitreo-Retinal Associates, Grand Rapids, Michigan
  - Retina Center, PA, Minneapolis, Minnesota
  - Mayo Clinic Department of Ophthalmology, Rochester, Minnesota
  - Barnes Retina Institute, St Louis, Missouri
  - Eyesight Ophthalmic Services, PA, Portsmouth, New Hampshire
  - The Institute of Ophthalmology and Visual Science (IOVS), Newark, New Jersey
  - Eye Associates of New Mexico, Albuquerque, New Mexico
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - The New York Eye and Ear Infirmary/Faculty Eye Practice, New York, New York
  - MaculaCare, New York, New York
  - Mount Sinai School of Medicine, Dept. of Ophthalmology, New York, New York
  - Retina Associates of Western New York, Rochester, New York
  - University of Rochester, Rochester, New York
  - Retina-Vitreous Surgeons of Central New York, PC, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - Western Carolina Retinal Associates, PA, Asheville, North Carolina
  - University of North Carolina, Chapel Hill, North Carolina
  - Charlotte Eye, Ear, Nose and Throat Assoc., PA, Charlotte, North Carolina
  - Wake Forest University Eye Center, Winston-Salem, North Carolina
  - Retina Associates of Cleveland, Inc., Beachwood, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - OSU Eye Physicians and Surgeons, LLC., Columbus, Ohio
  - Retina Vitreous Center, Edmond, Oklahoma
  - Dean A. McGee Eye Institute, Oklahoma City, Oklahoma
  - Retina Northwest, PC, Portland, Oregon
  - Casey Eye Institute, Portland, Oregon
  - Family Eye Group, Lancaster, Pennsylvania
  - University of Pennsylvania Scheie Eye Institute, Philadelphia, Pennsylvania
  - Retina Vitrous Consultants, Pittsburgh, Pennsylvania
  - Storm Eye Institute, Medical University of South Carolina, Charleston, South Carolina
  - Palmetto Retina Center, Columbia, South Carolina
  - Carolina Retina Center, Columbia, South Carolina
  - Southeastern Retina Associates, PC, Kingsport, Tennessee
  - Southeastern Retina Associates, P.C., Knoxville, Tennessee
  - Southwest Retina Specialists, Amarillo, Texas
  - Austin Retina Associates, Austin, Texas
  - Retina Research Center, Austin, Texas
  - Retina and Vitreous of Texas, Houston, Texas
  - Baylor Eye Physicians and Surgeons, Houston, Texas
  - Retina Consultants of Houston, PA, Houston, Texas
  - Texas Retina Associates, Lubbock, Texas
  - Valley Retina Institute, McAllen, Texas
  - Retinal Consultants of San Antonio, San Antonio, Texas
  - Retina Associates of Utah, P.C., Salt Lake City, Utah
  - Virginia Retina Center, Leesburg, Virginia
  - Retina Institute of Virginia, Richmond, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Spokane Eye Clinic, Spokane, Washington
  - University of Wisconsin-Madison, Dept of Ophthalmology/Retina Service, Madison, Wisconsin
  - Medical College of Wiconsin, Milwaukee, Wisconsin

REFERENCES:
- [Background] Wells JA, Glassman AR, Jampol LM, Aiello LP, Antoszyk AN, Baker CW, Bressler NM, Browning DJ, Connor CG, Elman MJ, Ferris FL, Friedman SM, Melia M, Pieramici DJ, Sun JK, Beck RW; Diabetic Retinopathy Clinical Research Network. Association of Baseline Visual Acuity and Retinal Thickness With 1-Year Efficacy of Aflibercept, Bevacizumab, and Ranibizumab for Diabetic Macular Edema. JAMA Ophthalmol. 2016 Feb;134(2):127-34. doi: 10.1001/jamaophthalmol.2015.4599. PMID 26605836
- [Background] Wells JA, Glassman AR, Ayala AR, Jampol LM, Bressler NM, Bressler SB, Brucker AJ, Ferris FL, Hampton GR, Jhaveri C, Melia M, Beck RW; Diabetic Retinopathy Clinical Research Network. Aflibercept, Bevacizumab, or Ranibizumab for Diabetic Macular Edema: Two-Year Results from a Comparative Effectiveness Randomized Clinical Trial. Ophthalmology. 2016 Jun;123(6):1351-9. doi: 10.1016/j.ophtha.2016.02.022. Epub 2016 Feb 27. PMID 26935357
- [Background] Jampol LM, Glassman AR, Bressler NM. Comparative Effectiveness Trial for Diabetic Macular Edema: Three Comparisons for the Price of 1 Study From the Diabetic Retinopathy Clinical Research Network. JAMA Ophthalmol. 2015 Sep;133(9):983-4. doi: 10.1001/jamaophthalmol.2015.1880. No abstract available. PMID 26087135
- [Background] Jampol LM, Glassman AR, Bressler NM, Wells JA, Ayala AR; Diabetic Retinopathy Clinical Research Network. Anti-Vascular Endothelial Growth Factor Comparative Effectiveness Trial for Diabetic Macular Edema: Additional Efficacy Post Hoc Analyses of a Randomized Clinical Trial. JAMA Ophthalmol. 2016 Dec 1;134(12):10.1001/jamaophthalmol.2016.3698. doi: 10.1001/jamaophthalmol.2016.3698. PMID 27711918
- [Background] Ross EL, Hutton DW, Stein JD, Bressler NM, Jampol LM, Glassman AR; Diabetic Retinopathy Clinical Research Network. Cost-effectiveness of Aflibercept, Bevacizumab, and Ranibizumab for Diabetic Macular Edema Treatment: Analysis From the Diabetic Retinopathy Clinical Research Network Comparative Effectiveness Trial. JAMA Ophthalmol. 2016 Aug 1;134(8):888-96. doi: 10.1001/jamaophthalmol.2016.1669. PMID 27280850
- [Background] Wells JA 3rd, Glassman AR, Jampol LM. Targeting the Effect of VEGF in Diabetic Macular Edema. N Engl J Med. 2015 Jul 30;373(5):481-2. doi: 10.1056/NEJMc1505684. No abstract available. PMID 26222565
- [Background] Bressler NM, Glassman AR, Hutton DW. Controversies in Using Off-Label Intravitreous Bevacizumab for Patients With Diabetic Macular Edema-Reply. JAMA Ophthalmol. 2017 Mar 1;135(3):291-292. doi: 10.1001/jamaophthalmol.2016.5686. No abstract available. PMID 28152135
- [Background] Bressler SB, Liu D, Glassman AR, Blodi BA, Castellarin AA, Jampol LM, Kaufman PL, Melia M, Singh H, Wells JA; Diabetic Retinopathy Clinical Research Network. Change in Diabetic Retinopathy Through 2 Years: Secondary Analysis of a Randomized Clinical Trial Comparing Aflibercept, Bevacizumab, and Ranibizumab. JAMA Ophthalmol. 2017 Jun 1;135(6):558-568. doi: 10.1001/jamaophthalmol.2017.0821. PMID 28448655
- [Background] Bressler NM, Beaulieu WT, Glassman AR, Blinder KJ, Bressler SB, Jampol LM, Melia M, Wells JA 3rd; Diabetic Retinopathy Clinical Research Network. Persistent Macular Thickening Following Intravitreous Aflibercept, Bevacizumab, or Ranibizumab for Central-Involved Diabetic Macular Edema With Vision Impairment: A Secondary Analysis of a Randomized Clinical Trial. JAMA Ophthalmol. 2018 Mar 1;136(3):257-269. doi: 10.1001/jamaophthalmol.2017.6565. PMID 29392288
- [Background] Glassman AR, Liu D, Jampol LM, Sun JK; Diabetic Retinopathy Clinical Research Network. Changes in Blood Pressure and Urine Albumin-Creatinine Ratio in a Randomized Clinical Trial Comparing Aflibercept, Bevacizumab, and Ranibizumab for Diabetic Macular Edema. Invest Ophthalmol Vis Sci. 2018 Mar 1;59(3):1199-1205. doi: 10.1167/iovs.17-22853. PMID 29625440
- [Background] Jampol LM, Glassman AR, Liu D, Aiello LP, Bressler NM, Duh EJ, Quaggin S, Wells JA, Wykoff CC; Diabetic Retinopathy Clinical Research Network. Plasma Vascular Endothelial Growth Factor Concentrations after Intravitreous Anti-Vascular Endothelial Growth Factor Therapy for Diabetic Macular Edema. Ophthalmology. 2018 Jul;125(7):1054-1063. doi: 10.1016/j.ophtha.2018.01.019. Epub 2018 Mar 7. PMID 29525602
- [Background] Bressler NM, Beaulieu WT, Maguire MG, Glassman AR, Blinder KJ, Bressler SB, Gonzalez VH, Jampol LM, Melia M, Sun JK, Wells JA 3rd; Diabetic Retinopathy Clinical Research Network. Early Response to Anti-Vascular Endothelial Growth Factor and Two-Year Outcomes Among Eyes With Diabetic Macular Edema in Protocol T. Am J Ophthalmol. 2018 Nov;195:93-100. doi: 10.1016/j.ajo.2018.07.030. Epub 2018 Aug 2. PMID 30077569
- [Background] Bressler SB, Odia I, Maguire MG, Dhoot DS, Glassman AR, Jampol LM, Marcus DM, Solomon SD, Sun JK; Diabetic Retinopathy Clinical Research Network. Factors Associated With Visual Acuity and Central Subfield Thickness Changes When Treating Diabetic Macular Edema With Anti-Vascular Endothelial Growth Factor Therapy: An Exploratory Analysis of the Protocol T Randomized Clinical Trial. JAMA Ophthalmol. 2019 Apr 1;137(4):382-389. doi: 10.1001/jamaophthalmol.2018.6786. PMID 30676635
- [Background] Bressler NM, Odia I, Maguire M, Glassman AR, Jampol LM, MacCumber MW, Shah C, Rosberger D, Sun JK; DRCR Retina Network. Association Between Change in Visual Acuity and Change in Central Subfield Thickness During Treatment of Diabetic Macular Edema in Participants Randomized to Aflibercept, Bevacizumab, or Ranibizumab: A Post Hoc Analysis of the Protocol T Randomized Clinical Trial. JAMA Ophthalmol. 2019 Sep 1;137(9):977-985. doi: 10.1001/jamaophthalmol.2019.1963. PMID 31246237
- [Background] Wells JA, Glassman AR, Ayala AR, Jampol LM. Reply. Ophthalmology. 2017 Jan;124(1):e5-e6. doi: 10.1016/j.ophtha.2016.04.032. No abstract available. PMID 27993277
- [Background] Wells JA, Glassman AR, Jampol LM, Ayala A, Bressler NM. Reply. Ophthalmology. 2017 Mar;124(3):e26-e27. doi: 10.1016/j.ophtha.2016.07.001. No abstract available. PMID 28219510
- [Background] Wells JA, Glassman AR, Bressler NM, Ayala AR, Jampol LM. Reply. Ophthalmology. 2017 Apr;124(4):e38-e39. doi: 10.1016/j.ophtha.2016.08.032. No abstract available. PMID 28335949
- [Background] Glassman AR, Duh EJ, Liu D, Jampol LM. Reply. Ophthalmology. 2018 Nov;125(11):e82. doi: 10.1016/j.ophtha.2018.05.004. No abstract available. PMID 30318048
- [Result] Diabetic Retinopathy Clinical Research Network; Wells JA, Glassman AR, Ayala AR, Jampol LM, Aiello LP, Antoszyk AN, Arnold-Bush B, Baker CW, Bressler NM, Browning DJ, Elman MJ, Ferris FL, Friedman SM, Melia M, Pieramici DJ, Sun JK, Beck RW. Aflibercept, bevacizumab, or ranibizumab for diabetic macular edema. N Engl J Med. 2015 Mar 26;372(13):1193-203. doi: 10.1056/NEJMoa1414264. Epub 2015 Feb 18. PMID 25692915
- [Derived] Talcott KE, Valentim CCS, Hill L, Stoilov I, Singh RP. Baseline Diabetic Retinopathy Severity and Time to Diabetic Macular Edema Resolution with Ranibizumab Treatment: A Meta-Analysis. Ophthalmol Retina. 2023 Jul;7(7):605-611. doi: 10.1016/j.oret.2023.02.003. Epub 2023 Feb 10. PMID 36774994
- [Derived] Pawloff M, Bogunovic H, Gruber A, Michl M, Riedl S, Schmidt-Erfurth U. SYSTEMATIC CORRELATION OF CENTRAL SUBFIELD THICKNESS WITH RETINAL FLUID VOLUMES QUANTIFIED BY DEEP LEARNING IN THE MAJOR EXUDATIVE MACULAR DISEASES. Retina. 2022 May 1;42(5):831-841. doi: 10.1097/IAE.0000000000003385. PMID 34934034
- [Derived] Roberts PK, Vogl WD, Gerendas BS, Glassman AR, Bogunovic H, Jampol LM, Schmidt-Erfurth UM. Quantification of Fluid Resolution and Visual Acuity Gain in Patients With Diabetic Macular Edema Using Deep Learning: A Post Hoc Analysis of a Randomized Clinical Trial. JAMA Ophthalmol. 2020 Sep 1;138(9):945-953. doi: 10.1001/jamaophthalmol.2020.2457. PMID 32722799

RESULTS

PARTICIPANT FLOW:
Groups:
- Ranibizumab: 0.3 mg intravitreal ranibizumab: Intravitreal injection of 0.3 mg ranibizumab at baseline and up to every 4 weeks using defined retreatment criteria.
Period: Overall Study
Arm/Group | Aflibercept | Bevacizumab | Ranibizumab
Started | 224 | 218 | 218
Completed | 208 | 206 | 206
Not Completed | 16 | 12 | 12
Not completed — Death | 3 | 5 | 3
Not completed — Withdrawal by Subject | 12 | 6 | 9
Not completed — Missed Visit | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aflibercept | Bevacizumab | Ranibizumab | Total
Number analyzed (Participants) | 224 | 218 | 218 | 660
Age, Customized [Mean (Standard Deviation); unit: years] | 60 (10) | 62 (10) | 60 (11) | 61 (10)
Sex/Gender, Customized [Number; unit: participants]
  Women | 110 | 103 | 94 | 307
  Men | 114 | 115 | 124 | 353
Race/Ethnicity, Customized [Number; unit: participants]
  White | 145 | 139 | 146 | 430
  Black/African American | 32 | 37 | 36 | 105
  Hispanic | 37 | 36 | 30 | 103
  Native Hawaiian/other Pacific Islander | 2 | 2 | 0 | 4
  American Indian/Alaskin Native | 1 | 0 | 0 | 1
  More than one race | 4 | 1 | 1 | 6
  Unknown/not reported | 1 | 1 | 1 | 3
  Asian | 2 | 2 | 4 | 8
Diabetes Type [Number; unit: participants]
  Type 1 | 22 | 12 | 16 | 50
  Type 2 | 196 | 205 | 196 | 597
  Uncertain | 6 | 1 | 6 | 13
Prior Myocardial Infarction [Number; unit: participants] | 13 | 14 | 16 | 43
Prior Coronary Artery Disease [Number; unit: participants] — Without myocardial infarction
  participants | 22 | 27 | 34 | 83
Prior Stroke [Number; unit: participants] | 8 | 13 | 10 | 31
Prior Transient Ischemic attacks [Number; unit: participants] | 6 | 8 | 10 | 24
Prior Hypertension [Number; unit: participants] | 177 | 181 | 175 | 533
Visual Acuity Letter Score [Median (Inter-Quartile Range); unit: units on a scale] — Best corrected visual acuity letter score as measured by a certified tester using an electronic visual acuity testing machine based on the Early Treatment Diabetic Retinopathy Study (ETDRS) method. Best value on the scale 97, worst 0.
  units on a scale | 69 [59 to 74] | 69 [60 to 72] | 68 [58 to 73] | 69 [59 to 73]
OCT Central Subfield [Median (Inter-Quartile Range); unit: Microns] — OCT = Optical Coherence Tomography
  Microns | 387 [310 to 483] | 376 [305 to 477] | 390 [310 to 493] | 387 [308 to 479]
Lens Status [Number; unit: participants]
  Phakic | 166 | 160 | 173 | 499
  Pseudophakic | 58 | 58 | 45 | 161
Diabetic Retinopathy Severity (ETDRS Level) [Number; unit: participants] — ETDRS = Early Treatment Diabetic Retinopathy Study; DR = diabetic retinopathy; PDR = proliferative diabetic retinopathy, NPDR = non-proliferative diabetic retinopathy, PRP = panretinal photocoagulation Criteria are based on the ETDRS fundus photographic risk factors for the progression of diabetic retinopathy. ETDRS report no. 12. Ophthalmology 1991; 98:823-833
  participants
    Absent of minimal NPDR | 7 | 6 | 5 | 18
    Mild to moderately severe NPDR | 150 | 131 | 145 | 426
    Severe NPDR | 17 | 15 | 18 | 50
    Prior PRP; without current PDR | 17 | 21 | 16 | 54
    Mild to moderate PDR | 28 | 31 | 23 | 82
    High risk PDR | 2 | 7 | 9 | 18
    Missing | 3 | 7 | 2 | 12
Prior Focal/Grid Laser for DME [Number; unit: participants] — DME = Diabetic macular edema Number of participants with prior focal/grid laser for DME in the study eye
  participants | 80 | 84 | 80 | 244
Prior Anti-VEGF for DME [Number; unit: participants] — VEGF = anti vascular endothelial growth factor DME = diabetic macular edema
  participants | 24 | 31 | 29 | 84
Prior other treatment for DME [Number; unit: participants] — DME = Diabetic macular edema
  participants | 14 | 12 | 11 | 37
Prior PRP [Number; unit: participants] — PRP = panretinal photocoagulation number of participants with prior panretinal photocoagulation in the study eye
  participants | 32 | 40 | 35 | 107

OUTCOME MEASURES:

1. Primary Outcome: Overall Change in Electronic Early Treatment Diabetic Retinopathy Study Visual Acuity Letter Score From Baseline to 1-year
Description: Visual Acuity was measured with the Electronic Early Treatment Study (E-ETDRS) visual acuity test. Unit of measure is based on the E-ETDRS letter score scale, 0-97, where 0 = worst and 97 = best.
Time Frame: Baseline to 1-year
Population: Visual acuity change truncated to +/- 3SD (-22 and +44) to minimize the effects of outliers for 6 eyes in the aflibercept group (4 on the positive end, 2 on the negative end) and 2 eyes in the bevacizumab group (both on the negative end).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aflibercept | Bevacizumab | Ranibizumab
Number analyzed (Participants) | 208 | 206 | 206
units on a scale | 13.3 (11.1) | 9.7 (10.1) | 11.2 (9.4)
Statistical Analysis 1: Comparison: Aflibercept vs Bevacizumab; Aflibercept vs. Bevacizumab; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 3.5, 95% CI 2-sided [1.4 to 5.7] — Reported P-values have been adjusted for multiple treatment group comparisons
Statistical Analysis 2: Comparison: Aflibercept vs Ranibizumab; Aflibercept vs. Ranibizumab; Test type: Superiority or Other; p = 0.034, ANCOVA; Mean Difference (Final Values) = 2.1, 95% CI 2-sided [0.1 to 4.2] — Reported P-values have been adjusted for multiple treatment group comparisons
Statistical Analysis 3: Comparison: Bevacizumab vs Ranibizumab; Ranibizumab vs. Bevacizumab; Test type: Superiority or Other; p = 0.12, ANCOVA; Mean Difference (Final Values) = 1.4, 95% CI 2-sided [-0.4 to 3.2] — Reported P-values have been adjusted for multiple treatment group comparisons

2. Secondary Outcome: Overall Change in Optical Coherence Tomography Central Subfield Thickness
Description: All baseline and 1-year optical coherence tomography (OCT) scans were graded by Duke Reading Center. In addition, a random sample of OCT images from other visits and images for which the investigator believed central grading was needed also were graded by Duke Reading Center.
  Baseline CSF values were converted from the thickness value measured on a Spectralis or Cirrus OCT machine to a Stratus equivalent value for 583 scans. One-year CSF values were converted from a thickness value measured on a Spectralis or Cirrus OCT machine to a Stratus equivalent value for 604 scans. When calculating change in CSF thickness, measurements taken on the same machine at both visits were not converted, since the conversion equation slope is nearly 1 and the constant difference does not affect the change calculation. Therefore, change in CSF thickness was calculated after converting either the baseline and/or follow-up thickness value from Spectralis or Cirrus to a Stratus equivalent value in 26 eyes.
Time Frame: baseline to 1-year
Population: In addition to participants missing the 1-year visit, 3 in the aflibercept group, 3 in the bevacizumab group, and 5 in the ranibizumab group had 1-year visits but unusable OCT data to compute change due to the scan being missing or ungradable at either baseline or 1 year.
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Aflibercept | Bevacizumab | Ranibizumab
Number analyzed (Participants) | 205 | 203 | 201
microns | -169 (138) | -101 (121) | -147 (137)
Statistical Analysis 1: Comparison: Aflibercept vs Bevacizumab; Aflibercept vs Bevacizumab; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -69.9, 95% CI 2-sided [-91.1 to -48.6] — Reported P-values have been adjusted for multiple treatment group comparisons
Statistical Analysis 2: Comparison: Aflibercept vs Ranibizumab; Aflibercept vs Ranibizumab; Test type: Superiority or Other; p = 0.036, ANCOVA; Mean Difference (Final Values) = -18.6, 95% CI 2-sided [-36 to -1.2] — Reported P-values have been adjusted for multiple treatment group comparisons
Statistical Analysis 3: Comparison: Bevacizumab vs Ranibizumab; Ranibizumab vs Bevacizumab; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -51.2, 95% CI 2-sided [-71.2 to -31.3] — Reported P-values have been adjusted for multiple treatment group comparisons

3. Primary Outcome: Change in Electronic Early Treatment Diabetic Retinopathy Study Visual Acuity Letter Score From Baseline to 1-year: Baseline Visual Acuity Letter Score <69
Description: as for outcome 1
Time Frame: Baseline to 1-year
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aflibercept | Bevacizumab | Ranibizumab
Number analyzed (Participants) | 102 | 102 | 101
units on a scale | 18.9 (11.5) | 11.8 (12.0) | 14.2 (10.6)
Statistical Analysis 1: Comparison: Aflibercept vs Bevacizumab; Aflibercept vs. Bevacizumab; Test type: Superiority or Other; p = 0.001, ANCOVA; Mean Difference (Final Values) = 6.5, 95% CI 2-sided [2.9 to 10.1] — Reported P-values have been adjusted for multiple treatment group comparisons
Statistical Analysis 2: Comparison: Aflibercept vs Ranibizumab; Aflibercept vs. Ranibizumab; Test type: Superiority or Other; p = 0.0031, ANCOVA; Mean Difference (Final Values) = 4.7, 95% CI 2-sided [1.4 to 8.0] — Reported P-values have been adjusted for multiple treatment group comparisons
Statistical Analysis 3: Comparison: Bevacizumab vs Ranibizumab; Ranibizumab vs Bevacizumab; Test type: Superiority or Other; p = 0.21, ANCOVA; Mean Difference (Final Values) = 1.8, 95% CI 2-sided [-1.1 to 4.8] — Reported P-values have been adjusted for multiple treatment group comparisons

4. Primary Outcome: Change in Electronic Early Treatment Diabetic Retinopathy Study Visual Acuity Letter Score From Baseline to 1-year: Baseline Visual Acuity Letter Score 78-69
Description: as for outcome 1
Time Frame: Baseline to 1-year
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aflibercept | Bevacizumab | Ranibizumab
Number analyzed (Participants) | 106 | 104 | 105
units on a scale | 8.0 (7.6) | 7.5 (7.4) | 8.3 (6.8)
Statistical Analysis 1: Comparison: Aflibercept vs Bevacizumab; Aflibercept vs Bevacizumab; Test type: Superiority or Other; p = 0.69, ANCOVA; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-1.3 to 2.7] — Reported P-values have been adjusted for multiple treatment group comparisons
Statistical Analysis 2: Comparison: Aflibercept vs Ranibizumab; Aflibercept vs Ranibizumab; Test type: Superiority or Other; p = 0.69, ANCOVA; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-2.3 to 1.5] — Reported P-values have been adjusted for multiple treatment group comparisons
Statistical Analysis 3: Comparison: Bevacizumab vs Ranibizumab; Ranibizumab vs Bevacizumab; Test type: Superiority or Other; p = 0.69, ANCOVA; Mean Difference (Final Values) = 1.1, 95% CI 2-sided [-0.9 to 3.1] — Reported P-values have been adjusted for multiple treatment group comparisons

5. Secondary Outcome: Change in Optical Coherence Tomography Central Subfield Thickness: Baseline Visual Acuity Letter Score <69
Description: as for outcome 2
Time Frame: baseline to 1-year
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Aflibercept | Bevacizumab | Ranibizumab
Number analyzed (Participants) | 101 | 100 | 99
microns | -210 (151) | -135 (152) | -176 (151)

6. Secondary Outcome: Change in Optical Coherence Tomography Central Subfield Thickness: Baseline Visual Acuity Letter Score 78-69
Description: as for outcome 2
Time Frame: baseline to 1-year
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Aflibercept | Bevacizumab | Ranibizumab
Number analyzed (Participants) | 104 | 103 | 102
microns | -129 (110) | -67 (65) | -119 (109)

7. Secondary Outcome: Overall Change in Retinal Volume
Description: Baseline volume values were converted from the thickness value measured on a Spectralis or Cirrus OCT machine to a Stratus equivalent value for 459 scans. One-year volume values were converted from a thickness value measured on a Spectralis or Cirrus OCT machine to a Stratus equivalent value for 472 scans. When calculating change in volume, measurements taken on the same machine at both visits were not converted, because the conversion equation slope is nearly 1 and the constant difference does not affect the change calculation. Therefore, change in volume was calculated after converting either the baseline and/or follow-up value from Spectralis or Cirrus to a Stratus equivalent value in 17 eyes.
Time Frame: Baseline to 1-year
Population: In addition to participants missing the 1-year visit, 46 in the aflibercept group, 53 in the bevacizumab group, and 44 in the ranibizumab group had 1-year visits but unusable OCT data to compute change due to the scan being missing or ungradable at either baseline or 1 year.
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Aflibercept | Bevacizumab | Ranibizumab
Number analyzed (Participants) | 162 | 153 | 162
mm^3 | -1.7 (1.6) | -1.0 (1.2) | -1.7 (1.5)

8. Secondary Outcome: Total Number of Injections Prior to 1 Year
Description: Only includes participants that completed the 1 year visit
Time Frame: Baseline to 1-year
Population: Seven study eyes received 1 injection and 2 eyes received 2 injections of 0.5 mg of ranibizumab prior to the FDA approving a 0.3 mg dosage of ranibizumab for diabetic macular edema treatment.
Measure: Mean (Standard Deviation); unit: Injections
Arm/Group | Aflibercept | Bevacizumab | Ranibizumab
Number analyzed (Participants) | 208 | 206 | 206
Injections | 9.2 (2.0) | 9.7 (2.3) | 9.4 (2.1)

9. Secondary Outcome: Total Number of Laser Treatments
Description: Only includes participants that completed the 1 year visit.
Time Frame: between 24 weeks and 1 year
Measure: Number; unit: participants
Arm/Group | Aflibercept | Bevacizumab | Ranibizumab
Number analyzed (Participants) | 208 | 206 | 206
participants
  0 | 132 | 91 | 111
  1 | 57 | 85 | 77
  2 | 19 | 30 | 18

10. Secondary Outcome: Eyes Receiving 1 or More Alternative Treatments for DME Other Than Laser
Time Frame: Baseline to 1-year
Measure: Number; unit: Eyes
Arm/Group | Aflibercept | Bevacizumab | Ranibizumab
Number analyzed (Participants) | 208 | 206 | 206
Eyes | 2 | 4 | 1

ADVERSE EVENTS:
Arm/Group | Aflibercept | Bevacizumab | Ranibizumab
Serious Adverse Events (participants affected / at risk) | 61/224 | 46/218 | 57/218
Other Adverse Events (participants affected / at risk) | 152/224 | 151/218 | 144/218
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aflibercept (N=224) | Bevacizumab (N=218) | Ranibizumab (N=218)
anaemia (Blood and lymphatic system disorders) | 3 | 0 | 1
anaemia of chronic disease (Blood and lymphatic system disorders) | 0 | 1 | 0
arrhythmia (Cardiac disorders) | 1 | 0 | 0
arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 2
Cardiac arrest (Cardiac disorders) | 1 | 1 | 0
cardiac failure (Cardiac disorders) | 0 | 1 | 2
cardiac failure congestive (Cardiac disorders) | 1 | 3 | 6
cardiomegaly (Cardiac disorders) | 1 | 0 | 0
coronary artery disease (Cardiac disorders) | 2 | 2 | 3
diastolic dysfunction (Cardiac disorders) | 1 | 0 | 0
hypertensive heart disease (Cardiac disorders) | 2 | 0 | 1
myocardial infarction (Cardiac disorders) | 3 | 1 | 3
palpitations (Cardiac disorders) | 0 | 0 | 1
pericardial effusion (Cardiac disorders) | 0 | 0 | 1
ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Diabetic ketoacidosis (Endocrine disorders) | 2 | 1 | 1
Glucocorticoid deficiency (Endocrine disorders) | 1 | 0 | 0
Hyperglycaemia (Endocrine disorders) | 1 | 0 | 0
Hypoglycaemia (Endocrine disorders) | 2 | 0 | 1
Cataract (Eye disorders) | 1 | 0 | 0
Endophthalmitis (Eye disorders) | 1 | 0 | 1
Glaucoma (Eye disorders) | 0 | 0 | 1
Visual acuity reduced (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 3 | 1
Clostridium difficile colitis (Gastrointestinal disorders) | 1 | 0 | 1
Colon cancer (Gastrointestinal disorders) | 0 | 1 | 1
Diabetic gastroparesis (Gastrointestinal disorders) | 2 | 0 | 1
Gastric cancer stage I (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 2 | 0
Gastroenteritis (Gastrointestinal disorders) | 0 | 1 | 1
Gastroenteritis viral (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal stoma complication (Gastrointestinal disorders) | 0 | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 3
Intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 5 | 4 | 1
Chest pain (General disorders) | 3 | 4 | 2
Death (General disorders) | 1 | 1 | 0
Device related infection (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 1 | 0
Pain (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1
Abscess (Infections and infestations) | 1 | 0 | 0
Escherichia infection (Infections and infestations) | 0 | 0 | 1
Infection (Infections and infestations) | 1 | 2 | 1
Influenza (Infections and infestations) | 1 | 0 | 0
Localised infection (Infections and infestations) | 2 | 2 | 3
Sepsis (Infections and infestations) | 3 | 1 | 1
Septic shock (Infections and infestations) | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subgaleal haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
International normalised ratio increased (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 2
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Obesity (Metabolism and nutrition disorders) | 1 | 0 | 0
Ankle fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Femur fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Inclusion body myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Lower limb fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Multiple fractures (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pelvic fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Upper limb fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Wrist fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Convulsion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Dizziness (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Dysarthria (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Encephalopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Headache (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Hypoaesthesia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Neuropathy peripheral (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Presyncope (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Somnolence (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Syncope (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
VIIth nerve paralysis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Vestibular neuronitis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 0 | 2
Mental disorder (Psychiatric disorders) | 1 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 1
Bladder prolapse (Renal and urinary disorders) | 0 | 0 | 1
Cystitis (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 4 | 6 | 9
Renal failure acute (Renal and urinary disorders) | 1 | 1 | 1
Renal failure chronic (Renal and urinary disorders) | 5 | 0 | 5
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0
Urinary tract infection (Renal and urinary disorders) | 3 | 1 | 0
Breast cancer (Reproductive system and breast disorders) | 0 | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Cardio-respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 6
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cellulitis (Skin and subcutaneous tissue disorders) | 2 | 6 | 2
Cellulitis gangrenous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 2 | 3
Furuncle (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 | 1 | 0
Foot amputation (Surgical and medical procedures) | 0 | 1 | 0
Gastric bypass (Surgical and medical procedures) | 1 | 0 | 0
Hip arthroplasty (Surgical and medical procedures) | 0 | 0 | 1
Stent placement (Surgical and medical procedures) | 0 | 2 | 0
Surgery (Surgical and medical procedures) | 1 | 0 | 2
Aortic stenosis (Vascular disorders) | 1 | 0 | 0
Arteriovenous fistula (Vascular disorders) | 1 | 0 | 1
Basilar artery occlusion (Vascular disorders) | 0 | 0 | 1
Cerebrovascular accident (Vascular disorders) | 0 | 1 | 3
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0
Haemorrhagic stroke (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 2 | 2 | 3
Hypotension (Vascular disorders) | 1 | 0 | 1
Ischaemic stroke (Vascular disorders) | 0 | 1 | 3
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 2 | 0 | 0
Transient ischaemic attack (Vascular disorders) | 0 | 1 | 2
Venous insufficiency (Vascular disorders) | 0 | 0 | 1
Venous stenosis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aflibercept (N=224) | Bevacizumab (N=218) | Ranibizumab (N=218)
Cataract (Eye disorders) | 14 (17) | 11 (14) | 14 (16)
Conjunctival haemorrhage (Eye disorders) | 30 (67) | 42 (83) | 25 (55)
Dry eye (Eye disorders) | 14 (23) | 9 (15) | 13 (18)
Eye irritation (Eye disorders) | 13 (28) | 16 (27) | 14 (24)
Eye pain (Eye disorders) | 27 (45) | 37 (50) | 21 (27)
Eye pruritus (Eye disorders) | 12 (15) | 10 (13) | 11 (20)
Lacrimation increased (Eye disorders) | 16 (22) | 7 (10) | 12 (14)
Vision blurred (Eye disorders) | 38 (55) | 39 (53) | 45 (77)
Visual acuity reduced (Eye disorders) | 18 (24) | 22 (27) | 17 (25)
Vitreous floaters (Eye disorders) | 41 (54) | 53 (70) | 37 (62)
Vitreous haemorrhage (Eye disorders) | 14 (17) | 18 (25) | 13 (15)
Headache (Nervous system disorders) | 15 (19) | 15 (19) | 15 (15)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 27 (31) | 20 (22) | 16 (17)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 12 (13) | 8 (8) | 13 (20)
Hypertension (Vascular disorders) | 24 (26) | 15 (16) | 23 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Trial results can not be discussed until they have been made available to the public.